CLINICAL TRIAL: NCT00809653
Title: Reducing the Pro-ischaemic Effects of Ambient Particulate Air Pollution in Patients With Coronary Heart Disease Using a Simple Face Mask Intervention
Brief Title: Reducing the Pro-ischaemic Effects of Air Pollution Exposure Using a Simple Face Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Professor David E Newby, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 167/2008/Patient
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2009-05

CONDITIONS: Angina Pectoris; Coronary Heart Disease; Blood Pressure; Heart Rate Variability
Keywords: Air pollution; Face mask; Myocardial ischaemia; Heart rate variability; Angina pectoris; Coronary heart disease
MeSH Terms: conditions — Angina Pectoris; Coronary Disease; Coronary Artery Disease | interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visit 1 (Experimental): 2 hour walk in city centre location in Beijing China
  Interventions: Device: No Face Mask
- Visit 2 (Experimental): 2 hour walk in city centre location in Beijing China
  Interventions: Device: Face Mask

INTERVENTIONS:
Device: No Face Mask — Subjects will not wear a face mask to reduce their personal air pollution exposure
  Arms: Visit 1
Device: Face Mask — Subjects will be asked to wear a simple face mask to reduce personal exposure to particulate air pollution. Subjects will be asked to wear the mask for 24 hours prior to the study day and the 24 hours of the study day. They will be instructed to wear the mask at all times when outdoors and as much as possible when indoors.
  Other Names: 3M Dust Respirator 8812
  Arms: Visit 2

SUMMARY:
Air pollution is a major cause of cardiorespiratory morbidity and mortality. The exact components of air pollution that underlie the cardiovascular effects are not yet known, but combustion-derived particulate matter is suspected to be the major cause. Epidemiological studies have shown that exposure to air pollution causes exacerbation of existing cardiorespiratory conditions leading to increased hospital admissions and death. The investigators have recently conducted a series of controlled exposure studies to urban particulate matter and diesel exhaust in healthy volunteers and patients with coronary heart disease. The investigators found that controlled exposure to dilute diesel exhaust in patients with prior myocardial infarction induced asymptomatic myocardial ischaemia with an increase in electrocardiographic measures of myocardial ischaemia. Whilst important, further questions remain: (i) does air pollution exposure exacerbate ischaemia and reduce exercise tolerance in patients with symptomatic angina pectoris, (ii) do "real world" exposures as encountered in the urban environment of major cities have similar effects, and (iii) can a simple face mask intervention to reduce exposure to particulate air pollution improve health outcomes in patients with coronary heart disease?

DETAILED DESCRIPTION:
100 patients with stable angina pectoris will be recruited from the HPS-THRIVE cohort or from the cardiology outpatient department at the Fuwai Hospital in Beijing. Patients will attend the department first thing in the morning on two occasions, separated by at least 1 week. All subjects will be fitted with a 12-lead Holter monitor and 24-hour ambulatory blood pressure monitor. They will be issued with a diary to record their activities and symptoms.

Patients will be randomised to wear a simple facemask for one of their visits (3M Dust Respirator 8812). When randomised to wear a mask, subjects will be asked to wear the mask as much as possible in the 24 hours prior to the study day and for the 24 hours of the study day (48 hours in total). Subjects will be instructed to wear the mask at all times when outdoors, and as much as possible when indoors.

On both visits, patients will be asked to walk along a prespecified route for 2 hours in a city centre location in Beijing. During this period patients will walk at their own pace for 15 mins and rest for 5 mins for a total of 120 mins (6 cycles). After the walk, subjects will return to the department and the pollution equipment switched off. A formal BRUCE protocol exercise stress test will be performed as soon as possible after finishing the 2-hour walk, and blood tests will be taken just prior to the exercise stress test (10-20mls in total). Subjects will be asked to wear the ambulatory blood pressure monitor and the Holter ECG monitor for a total of 24 hours, returning the following day to have this removed. Personal exposure to air pollution will be determined during the 2 hour walk with a series of monitors contained within a small backpack.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary heart disease
* Symptoms of angina pectoris
* Evidence of coronary heart disease by angiography or by exercise stress testing

Exclusion Criteria:

* Current smokers
* History of arrhythmia
* Severe 3 vessel coronary heart disease or left main stem stenosis that has not been revascularised
* Resting conduction abnormality
* Digoxin therapy
* Uncontrolled hypertension
* Renal failure
* Hepatic failure
* Acute coronary syndrome or unstable symptoms within 3 months
* Significant occupation exposure to air pollution

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Myocardial ischaemic burden determined using continuous electrographic monitoring | During 2 hour walk and subsequent 24 hour period

SECONDARY OUTCOMES:
Symptoms of angina pectoris assessed by patient diary and GTN use | During 2 hour walk and subsequent 24 hour period
Biochemical markers of myocardial ischaemia | After 2 hour city centre walk
Systemic inflammatory markers | After 2 hour city centre walk
Blood pressure | During 2 hour walk and for subsequent 24 hours
Heart rate and heart rate variability | During 2 hour walk and subsequent 24 hour period
Personal exposure to air pollutants | During 2 hour walk
Exercise capacity, time to symptoms and time to 1mm ST segment depression on standard treadmill exercise testing | Immediately after 2 hour city centre walk

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, MD, Principal Investigator — Chinese Academy of Medical Sciences and Peking Medical Union College; David E Newby, PhD FRCP, Principal Investigator — University of Edinburgh
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Medical Union College, Beijing, China

REFERENCES:
- [Background] Mills NL, Tornqvist H, Gonzalez MC, Vink E, Robinson SD, Soderberg S, Boon NA, Donaldson K, Sandstrom T, Blomberg A, Newby DE. Ischemic and thrombotic effects of dilute diesel-exhaust inhalation in men with coronary heart disease. N Engl J Med. 2007 Sep 13;357(11):1075-82. doi: 10.1056/NEJMoa066314. PMID 17855668
- [Derived] Langrish JP, Watts SJ, Hunter AJ, Shah AS, Bosson JA, Unosson J, Barath S, Lundback M, Cassee FR, Donaldson K, Sandstrom T, Blomberg A, Newby DE, Mills NL. Controlled exposures to air pollutants and risk of cardiac arrhythmia. Environ Health Perspect. 2014 Jul;122(7):747-53. doi: 10.1289/ehp.1307337. Epub 2014 Mar 25. PMID 24667535
- [Derived] Langrish JP, Li X, Wang S, Lee MM, Barnes GD, Miller MR, Cassee FR, Boon NA, Donaldson K, Li J, Li L, Mills NL, Newby DE, Jiang L. Reducing personal exposure to particulate air pollution improves cardiovascular health in patients with coronary heart disease. Environ Health Perspect. 2012 Mar;120(3):367-72. doi: 10.1289/ehp.1103898. PMID 22389220